CLINICAL TRIAL: NCT04279301
Title: Causes and Outcomes of Neonatal Admission in Neonatal Intensive Care Unit of Assuit University Children Hospital(AUCH)
Brief Title: Neonatal Admission in Assuit University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Naguib Khairy, Principle Investigator, Assiut University
Other Study IDs: Neonatal admission in AUCH
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Neonatal Disease
Keywords: Neonatal morbidity
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are many causes of admission of neonates in Neonatal Intensive Care Unit.So knowing such causes and their outcomes will give us knowledge about different risk factors of each disease and the prognosis of each cause.

DETAILED DESCRIPTION:
The rapid decline in neonatal mortality during the past 4 decades has been attributed to improvements in neonatal intensive care. This decline was attributable to improved condition of the infants on NICU(Neonatal Intensive Care Unit) admission (improved birth weight, higher Apgar scores, and better physiologic ability).

There are multiple risk factors related to admission of newborns at NICU as low birth weight , neonatal sepsis , hypothermia , hypoglycemia , respiratory distress and other factors. These risk factors are also considered as causes of death beside prematurity and congenital malformations.

One of the most important risk factors for admission and is considered as a major cause of death is premature infants. Neonatal intensive care has become a cornerstone for treatment of premature infants worldwide.

Another group is low birth weight (LBW) infants. LBW babies face increased risk of a myriad of physical and developmental problems. Before the era of neonatal intensive care units, few VLBW infants survived. Today, babies who weigh as little as a pound and developed in the uterus for as early as 26 weeks have been known to survive. LBW babies need high cost of intensive neonatal care and adequate nursing coverage.

Neonatal respiratory morbidity in term infants is another cause of admission and death in neonates and is multifactorial in aetiology.

Neonatal sepsis as well is one of the most common reasons for admission to neonatal units in developing countries. It is also a major cause of mortality in both developed and developing countries.

Hypoglycaemia also plays an important role as it accounts for approximately one-tenth of term admissions to neonatal units can cause long-term neurodevelopmental impairment and is associated with the significant burden to the affected infants, families and the health system.

Knowing the disease patterns and causes in the neonatology unit and the disease-wise outcome can inform the required efforts to reduce morbidity and mortality. Thus, in this study we will assess the causes and risk factors for neonatal admission at NICU of Assuit University Children Hospital (AUCH) and the outcome of them.

ELIGIBILITY:
Inclusion Criteria:

* All neonates delivered in Assuit University Hospital and admitted at NICU of Assuit University Children Hospital.

Exclusion Criteria:

* Patients delivered outside Assuit University Hospital.
* Patients with missing diagnosis or died before reaching diagnosis.
* Patients with missing clinical outcomes.
* Patients admitted for observation and discharged at the same day of admission.

Ages: 1 Hour to 1 Month | Sex: All
Age Groups: Child
Study Population: Neonates delivered in Assuit University Hospital and need admission in neonatology unit of Assuit University Children Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Detection of cause of admission of neonate in Neonatology Unit and the outcome of this cause | baseline
  Analysis of these causes and their outcomes

REFERENCES:
- [Background] Seid SS, Ibro SA, Ahmed AA, Olani Akuma A, Reta EY, Haso TK, Fata GA. Causes and factors associated with neonatal mortality in Neonatal Intensive Care Unit (NICU) of Jimma University Medical Center, Jimma, South West Ethiopia. Pediatric Health Med Ther. 2019 May 3;10:39-48. doi: 10.2147/PHMT.S197280. eCollection 2019. PMID 31191085
- [Background] Quinn CE, Sivasubramaniam P, Blevins M, Al Hajajra A, Znait AT, Khuri-Bulos N, Faouri S, Halasa N. Risk factors for neonatal intensive care unit admission in Amman, Jordan. East Mediterr Health J. 2016 Jun 15;22(3):163-74. doi: 10.26719/2016.22.3.163. PMID 27334073
- [Background] Goswami IR, Ghosh JK, Sinha MK, Begum H, Chatterjee S. Can the special care neonatal unit admission cut-off be lowered down to 1500g babies? Indian J Pediatr. 2009 Sep;76(9):937-9. doi: 10.1007/s12098-009-0185-z. Epub 2009 Nov 4. PMID 19904507
- [Background] Alkiaat A, Hutchinson M, Jacques A, Sharp MJ, Dickinson JE. Evaluation of the frequency and obstetric risk factors associated with term neonatal admissions to special care units. Aust N Z J Obstet Gynaecol. 2013 Jun;53(3):277-82. doi: 10.1111/ajo.12070. Epub 2013 Mar 13. PMID 23731095
- [Background] Quddus AR, Islam MN, Uddin MB, Mahmud AA, Badruzzaman M, Saha SK, Sattar S, Afreen KF. Study of Risk Factors, Causative Organisms & Their Sensitivity Pattern in Neonatal Sepsis in a Community Based Tertiary Level Hospital. Mymensingh Med J. 2019 Oct;28(4):839-848. PMID 31599249
- [Background] Dassios T, Greenough A, Leontiadi S, Hickey A, Kametas NA. Admissions for hypoglycaemia after 35 weeks of gestation: perinatal predictors of cost of stay. J Matern Fetal Neonatal Med. 2019 Feb;32(3):448-454. doi: 10.1080/14767058.2017.1381905. Epub 2018 Jan 31. PMID 28922987